CLINICAL TRIAL: NCT02472366
Title: A Non-Randomized, Open-Label, Single Center Phase 4 Study of the Effect and Safety of ILUVIEN® in Chronic Diabetic Macular Edema Patients Considered Insufficiently Responsive to Available Therapies (Laser, Anti-VEGF) With or Without Intravitreal Corticosteroid Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alimera Sciences (Industry)
Responsible Party: Sponsor
Organization: ANI Pharmaceuticals (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M-01-13-002
Record Dates: First submitted 2015-06-10; First posted 2015-06-15 (Estimated); Results first posted 2015-09-16 (Estimated); Last update posted 2015-09-16 (Estimated); Status verified 2015-08

CONDITIONS: Chronic Diabetic Macular Edema
MeSH Terms: interventions — Fluocinolone Acetonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- laser (Other): laser with or without prior history of intraocular corticosteroid therapy
  Interventions: Drug: ILUVIEN
- laser and anti-VEGF (Other): laser and anti-VEGF therapy with or without prior history of intraocular corticosteroid therapy
  Interventions: Drug: ILUVIEN

INTERVENTIONS:
Drug: ILUVIEN

SUMMARY:
A phase 4 trial evaluating the effect and safety of ILUVIEN in chronic DME patients insufficiently responsive to available therapies.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥18 years of age, of either sex that have signed informed consent / been well informed by the treating physician.
2. DME based on investigator's clinical evaluation and demonstrated using fundoscopic photography and spectral domain OCT.
3. Mean central foveal thickness (central subfield thickness) ≥350 microns in the study eye as measured using spectral domain OCT.
4. Vision impairment (20/60 to 20/400 using Snellen visual acuity equivalent) related to DME.
5. Previous treatment in the study eye with laser photocoagulation for DME, including focal/grid and pan-retinal, at least 3 months prior to the screening visit and ≥3 monthly anti-VEGF treatments (group 1).
6. Previous treatment in the study eye with laser photocoagulation for DME at least 3 months prior to the screening visit (group 2) and treatment with an intraocular anti-VEGF therapy not possible.
7. Patients considered as insufficiently responsive to prior therapy for DME, as defined by the study physician.

Exclusion Criteria:

1. IOP >21 mmHg at screening in the study eye.
2. Historical rise in IOP >25 mmHg following treatment with an intravitreal corticosteroid in the study eye.
3. Use of ≥2 IOP-lowering medications to control IOP at screening in the study eye.
4. Patients that have vitreomacular traction in DME and opaque media in the study eye.
5. Patients with severe proliferative diabetic retinopathy requiring pan retinal photocoagulation in the study eye.
6. Pregnant or breastfeeding.
7. Patients diagnosed with active angiographic central vein ischaemia prior to screening in the study eye.
8. Patients that have received pan retinal photocoagulation or undergone cataract surgery in the 3 months prior to the study start date in the study eye.
9. Patients with contraindications according to the current SPC:

   1. The presence of pre-existing glaucoma.
   2. Active or suspected ocular or periocular infection.
   3. The patient is hypersensitive to the active agent or to one of the excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-01; Primary Completion 2015-03 (Actual); Study Completion 2015-05 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Laser: laser with or without prior history of intraocular corticosteroid therapy
  ILUVIEN
- Laser and Anti-VEGF: laser and anti-VEGF therapy with or without prior history of intraocular corticosteroid therapy
  ILUVIEN
Period: Overall Study
Arm/Group | Laser | Laser and Anti-VEGF
Started | 6 (6 subjects receiving ILUVIEN, 7 eyes receiving ILUVIEN) | 10
Completed | 5 | 10
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Laser | Laser and Anti-VEGF | Total
Number analyzed (Participants) | 6 | 10 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.65 (9.014) | 60.87 (11.006) | 63.04 (10.398)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 7
  Male | 4 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: Changes in Best Corrected Visual Acuity From Baseline
Description: Best Corrected Visual Acuity is measured using an ETDRS eye chart and is reported as the number of letters read correctly in the study and/or fellow eye.
Time Frame: Change from Baseline to 12 months post ILUVIEN administration
Population: For the "Laser" arm group, 6 patients were enrolled and 7 eyes were treated with ILUVIEN
Measure: Mean (Standard Deviation); unit: Best Corrected VA Letter Score
Units Other Than Participants: Eyes
Arm/Group | Laser | Laser and Anti-VEGF
Number analyzed (Participants) | 6 | 10
Number analyzed (Eyes) | 7 | 10
Best Corrected VA Letter Score | 3.5 (7.40) | 0.9 (15.79)

2. Secondary Outcome: Changes in Intraocular Pressure (IOP)
Time Frame: Change from Baseline to 12 months post ILUVIEN administration
Population: for "laser" arm group, 6 patients enrolled with 7 eyes receiving ILUVIEN
Measure: Mean (Standard Deviation); unit: mmHg
Units Other Than Participants: Eyes
Arm/Group | Laser | Laser and Anti-VEGF
Number analyzed (Participants) | 6 | 10
Number analyzed (Eyes) | 7 | 10
mmHg | 1.7 (1.86) | 2.9 (6.28)

3. Secondary Outcome: Changes in Central Subfield Thickness
Time Frame: Change from Baseline to 12 months post ILUVIEN administration
Population: For "Laser" arm group, there were 6 patients enrolled but 7 eyes treated
Measure: Mean (Standard Deviation); unit: microns
Units Other Than Participants: Eyes
Arm/Group | Laser | Laser and Anti-VEGF
Number analyzed (Participants) | 6 | 10
Number analyzed (Eyes) | 7 | 10
microns | -362.2 (130.59) | -251.3 (268.29)

4. Secondary Outcome: Changes in Macular Volume
Time Frame: Change from Baseline to 12 months post ILUVIEN administration
Population: For "laser" arm group, 6 patients were enrolled with 7 eyes receiving ILUVIEN
Measure: Mean (Standard Deviation); unit: mm^3
Units Other Than Participants: Eyes
Arm/Group | Laser | Laser and Anti-VEGF
Number analyzed (Participants) | 6 | 10
Number analyzed (Eyes) | 7 | 10
mm^3 | -1.610 (1.1979) | -1.137 (3.4345)

5. Post Hoc Outcome: Change in Best Corrected Visual Acuity From Baseline
Description: A subgroup analysis was performed in which only pseudophakic subjects were included. Best Corrected Visual Acuity is measured using an ETDRS eye chart and is reported as the number of letters read correctly in the study and/or fellow eye.
Time Frame: Change from Baseline to 12 months post ILUVIEN administration
Population: For the "Laser" arm group, 6 patients were enrolled and 7 eyes were treated with ILUVIEN
Measure: Mean (Standard Deviation); unit: Best Corrected VA Letter Score
Units Other Than Participants: Eyes
Arm/Group | Laser | Laser and Anti-VEGF
Number analyzed (Participants) | 6 | 5
Number analyzed (Eyes) | 7 | 5
Best Corrected VA Letter Score | 5.6 (8.70) | 9.4 (11.46)

ADVERSE EVENTS:
Time Frame: The safety and tolerability of ILUVIEN was monitored over 12 months.
Arm/Group | Laser | Laser and Anti-VEGF
Serious Adverse Events (participants affected / at risk) | 0/6 | 2/10
Other Adverse Events (participants affected / at risk) | 2/6 | 3/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Laser (N=6) | Laser and Anti-VEGF (N=10)
Stroke (Nervous system disorders) | 0 (0) | 1 (1)
Cataract Surgery (Surgical and medical procedures) | 0 (0) | 1 (2)
Vitrectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Laser (N=6) | Laser and Anti-VEGF (N=10)
Intra-ocular pressure (30 mmHg) (Eye disorders) | 1 (1) | 0 (0)
Dislocated Shoulder (General disorders) | 1 (1) | 0 (0)
Intra-ocular pressure (25mmHG) (Eye disorders) | 0 (0) | 2 (2) — 1 event occurred in the fellow eye
Intra-ocular pressure (28mmHg) (Eye disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less